CLINICAL TRIAL: NCT04841876
Title: Sports-related Concussion: Physiological, Biomechanical and Cognitive Methodology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Prof Baker Julien, Professor, Hong Kong Baptist University
Other Study IDs: REC/20-21/0452
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Concussion (Diagnosis)
Keywords: Blood-based biomarkers; Motor control; Cognitive function Skill; Biomechanics; Sport-related concussion
MeSH Terms: conditions — Brain Concussion; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-1: Participants who are professional rugby-7s plays will be randomly assigned to one of the two groups. For Group-1, participants will be asked to play three consecutive rugby matches, with 40 min for each match. The total duration will be 2 hours. There is no additional intervention on this group.
  Interventions: Other: rugby matches
- Group 2: Participants who are professional rugby-7s plays will be randomly assigned to one of the two groups. For Group-2, participants will be asked to only watch the rugby matches. They will not received any intervention.

INTERVENTIONS:
Other: rugby matches — standard rugby-7s match
  Groups: Group-1

SUMMARY:
The study aims to investigate the changes in physiological, biomechanical and cognitive performance under a traumatic sport-event (i.e., rugby match).

DETAILED DESCRIPTION:
Background: Regular participation in moderate-to-vigorous physical activity in contact sports may be related to increases in cerebrovascular injury and head trauma. The diagnosis of head injury is lacking in validated objective measures immediate post event. Diagnostic markers may also be confounded by the exercise type and intensity. Therefore, it deserves further examination on a variety of functional (biomechanical and motor control) performance and blood-based biomarkers to determine how these indicators are affected by contact sport and the incidence of head injury. The study aims to investigate the changes in physiological, biomechanical and cognitive performance under a traumatic sport-event.

Methods: The study will use a two-group randomized controlled trial (RCT) with double-blinded approach, comprising a traumatic sport-event group and a control group. Thirty rugby-7s players will be recruited and randomly assigned to one of the two groups, where the intervention group will play three consecutive rugby matches. Data will be collected pre and post rugby match performance. Particularly, demographic and anthropometric data will be collected at baseline and pre-match. Venous blood, biomechanical data, and cognitive-motor task data will be collected at baseline, pre-match, and after each of 3 consecutive matches. Notational analysis will be performed after each match. Venous blood will be collected 24, 48, and 72 hours after the 3rd match.

Discussion: It is expected to see a reduction in whole-body movement, coordination, and cognitive-motor tasks as the number of games continues through fatigue and/or traumatic events. It is also expected that changes in blood-based biomarker concentrations to correlate with changes in biomechanical and cognitive-motor tasks. The proposed study will yield meaningful, ecologically valid research regarding the occurrence of concussive events, the influence of these on the biological system of the performer, with direct impact on clinicians, scientists, and sport governing bodies. The scope of this study will have implications on health and wellbeing within sporting populations at all levels, genders, and ages. Additionally, the findings will facilitate greater understanding about the human responses to exercise induced trauma.

ELIGIBILITY:
Inclusion Criteria:

(1) Participants should be 18 years old or above; (2) no restriction of physical mobility; (3) no uncontrollable mental disorders; and (4) professional rugby-7s player.

Exclusion Criteria:

(1) less than 18 years old; (2) have restriction of physical mobility; (3) have uncontrollable mental disorders; and (4) training duration of rugby is less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be the professional rugby-7s players at the Hong Kong Sports Institute (Sha Tin, N.T. Hong Kong, China).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood indicator | Data will be collected at pre-match, and after each of 3 consecutive matches, and 24-, 48-, and 72-hours post-match
  The day before tournament play each participant will donate 10mL of blood into two separate 5 mL serum separation vacutainer tubes (SST)s (Becton Dickinson, Rutherford, NJ, USA) On the day of the tournament another 10 mL blood sample will be collected into two separate 5 mL SSTs before the first rugby match and then immediately after each successive rugby match. After the last rugby match, blood will be drawn immediately after as well as 24-, 48-, and 72-hours post-match into two separate 5 mL SSTs.
  All blood draws will be performed using the standard venepuncture method. After blood is collected in the SSTs it will be allowed to clot for one hour at room temperature. Following the incubation period, the SSTs will be centrifuged at 1250 g for 10 min at 4°C. Once centrifugation is complete the serum supernatant will be removed and placed into two tubes (Eppendorf®) and stored at -80°C until analysis.
Change in biomechanical performance: Throwing task | Data will be collected at pre-match, and after each of 3 consecutive matches
  During the ecologically valid movement task participants will perform an anticipated and unanticipated passing drill where the player runs and passes with maximum speed to a target. Participants will be labelled using a modified full body 6DOF kinematic model, 38 retroreflective markers (14 mm in diameter) will be affixed to the skin using double sided tape. Synchronised Three-dimensional kinematic (14 camera, Vicon Vantage Oxford Metrics, Oxford, UK, 250 Hz) and kinetic data (force plates: four 600mm x 900 mm Kistler 9287BA, Winterhur, Switzerland) will be collected.
Change in biomechanical performance: mBESS | Data will be collected at pre-match, and after each of 3 consecutive matches
  During the mBESS test participants will be instructed to stand on their non-dominant foot with dominant leg held with 30° hip flexion, 45° knee flexion and in tandem stance with eyes closed and hands placed on the iliac crest for 30 seconds. Shoes will be left on. Participants will stand on a force plate within the capture area.
Change in biomechanical performance: Tandem Gait | Data will be collected at pre-match, and after each of 3 consecutive matches.
  Participants will be instructed to stand with their feet together behind a starting line with shoes on. Participants will walk heel-to-toe, so that toes of one foot touch the heel of the next at each step to complete a 3m walk (eyes open) as quickly and accurately as possible, turning 180° and returning (total 6m). A 38mm wide (sports tape), 3 metre line will mark the walkway on the floor. If participants step off the line, have a separation between their heel and toe, or touch or grab the examiner or an object they will be corrected and asked to continue.
Change in biomechanical performance: Finger-to-nose | Data will be collected at pre-match, and after each of 3 consecutive matches.
  In line with a modified SCAT 5 protocol, finger to nose task will be performed within the data capture area with the participant standing with both feet on the force plate. Instructions will be delivered as follows: "I am going to test your coordination now. Stand on both feet with eyes open and your dominant arm outstretched in front of you. On the start signal, perform five successive finger to nose repetitions using your index finger to touch the tip of the nose, and then return to the starting position. Perform the movements as quickly and as accurately as possible."
Change in cognitive-motor performance: Purdue Pegboard | Data will be collected at pre-match, and after each of 3 consecutive matches.
  Perdue pegboard was used to explore bimanual finger and hand dexterity (Tiffin, 1968; Tiffin & Asher, 1948). The Purdue Pegboard consists of two parallel rows of 25 holes, in which pegs initially located in two laterally located cups, are inserted, followed by collars and washers are initially positioned in two middle cups. Four sub-tests are performed. In the first sub-test, as many pins as possible are placed in the holes (from top to bottom), first with the preferred hand, then in the second sub-test with the non-preferred hand, and in the third sub-test with both hands, within a 30-s time period. In the fourth subtest, the participant uses both hands alternately to construct "assemblies," consisting of a peg, a washer, a collar, and another washer within 1 minute.
Change in cognitive-motor performance: Tapping Task | Data will be collected at pre-match, and after each of 3 consecutive matches.
  The finger-tapping test (FTT) examines motor speed and lateralized coordination. To run the test, the palm should will be taped to a flat board, with fingers extended. The index finger will then 'tap' on a computer key board button. Participants will be asked to tap each finger as quickly as possible on the button over a 10-s time period. Three trials with each finger will be run. Number of taps will be averaged across trials, in order to increase the number on the counting device with each tap. https://link.springer.com/referenceworkentry/10.1007/978-1-4419-1698-3_343
Change in cognitive-motor performance: Stroop word test | Data will be collected at pre-match, and after each of 3 consecutive matches.
  The Stroop colour test will be performed on a computer using the online demo test: https://www.psytoolkit.org/experiment-library/stroop.html. Participants will sit comfortably at the computer workstation and be shown a demonstration of how to perform the test. After which, the 2-minute demo test will be completed. Stroop will be run with verbal response and with keyboard response. 40 words will be presented for 2 seconds each, and the four colours red, blue, green and yellow used. For the verbal response a screen+camera recording will be used to record the Stroop word and the participant response, to allow scoring after the test is completed.
Change in cognitive-motor performance: Reaction time | Data will be collected at pre-match, and after each of 3 consecutive matches.
  A digital reaction time test will be used to quantify reaction time. The test https://humanbenchmark.com/tests/reactiontime will be performed 5 times with each hand.
Change in cognitive-motor performance: Working memory | Data will be collected at pre-match, and after each of 3 consecutive matches.
  Digit Span Backward test, participants are presented with a series of digits to be repeated backward. As detailed by Ramsay and Reynold (1995) the score of working memory is calculated from the temporal responses to the increasing number strings. The raw score will be used as a measure of working memory.

SECONDARY OUTCOMES:
Demographics and anthropometrics | At baseline
  At baseline, a series of demographic information and covariates related to sport concussion will be collected, including age, sex, duration of training, medication use, medical history (e.g., mental health problems), health behaviours (e.g., exercise prior to blood draw, alcohol consumption, smoking), history of rugby play, rugby position, and concussion history.
  In addition to standing height and total body mass, personalised anthropometric measures will be calculated for each rugby player using digitised coordinate data from whole-body static images, these measures will provide body segment inertia characteristics based on (Gittoes et al., 2009, and Yeadon, 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Julien S. Baker, Ph.D., D.Sc., Principal Investigator — Hong Kong Baptist University

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, statistical plan, informed consent form, and research output.